CLINICAL TRIAL: NCT07400029
Title: A Phase II Trial of Obecabtagene Autoleucel Consolidation in Adult Patients With Acute Lymphoblastic Leukemia in First Complete Remission Without Measurable Residual Disease
Brief Title: A Study of Obecabtagene Autoleucel in People With B-cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-342
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Obecabtagene Autoleucel; B-cell; 25-342
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): will enroll Philadelphia chromosome negative patients
  Interventions: Drug: Obecabtagene Autoleucel
- Cohort B (Experimental): is an exploratory cohort that will enroll Philadelphia chromosome positive patients
  Interventions: Drug: Obecabtagene Autoleucel

INTERVENTIONS:
Drug: Obecabtagene Autoleucel — given as infusion

SUMMARY:
The researchers are doing this study to find out whether obecabtagene autoleucel (obe-cel) is an effective treatment for people with B-cell acute lymphoblastic leukemia (ALL) that is in complete remission (CR, meaning all signs of cancer are gone) with no measurable residual disease (MRD-negative, meaning there are no detectable cancer cells). Participants in this study will have received past treatment for their B-cell ALL, and their disease will be in MRD-negative CR for the first time (first MRD-negative CR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD19+ B-cell ALL.

  * Both Ph-negative and Ph-positive are allowed
  * Patients with EMD must have detectable disease in the bone marrow (by flow cytometry or molecular methods) in order to follow MRD.
* Patients aged ≥ 40 years at time of screening A.
* Patients aged 30-39 years (at time of Screening A) are allowed in the presence of high-risk comorbidities or poor tolerability of chemotherapy (e.g. history or experienced pancreatitis with therapy, BMI ≥40kg/m2, underlying liver disease precluding safer administration of pediatric inspired regimens, any further combination of documented severe comorbidities that the investigator judges to be incompatible with administering an intensive pediatric or pediatric-inspired standard chemotherapy regimen).
* In MRD negative CR or CR with incomplete hematologic recovery (CRi) at the time of screening. MRD will be assessed by flow cytometry and/or molecular testing such as ClonoSEQ at the minimum sensitivity of 10-4 from the bone marrow. Patients with MRD <10^-4 will be eligible.
* Patients may receive more than one course of upfront induction and/or consolidation, but must be in MRD- CR/CRi at time of screening, within 4 months from initiation of treatment. The 4-month window will be measured from the first day of anti-leukemic therapy initiation (excluding steroid prophase) until the Screening A test for the trial.

Frontline regimens include but are not limited to:

* HyperCVAD or mini-hyper-CVD
* Asparaginase-containing multiagent chemotherapy (e.g. CALGB10403, pediatric inspired chemo)
* Inotuzumab or blinatumomab with or without chemotherapy
* Tyrosine kinase inhibitor plus steroids, chemotherapy, or blinatumomab

  - Adequate organ function at time of screening A, including:
* ALT or AST ≤5x ULN and total bilirubin ≤2 (or ≤3 if history of Gilbert's syndrome or leukemic infiltration of the liver)
* Serum creatinine <2.0mg/dL
* SaO2 ≥92% on room air
* Left ventricular ejection fraction (LVEF) ≥50% within 1 month of screening

  * ECOG performance status 0-2
  * CD19 expression is required at any time since diagnosis. CD19 expression may be detected by immunohistochemistry or by flow cytometry. Patients receiving prior blinatumomab are eligible if there is no documentation of CD19-negative disease after blinatumomab.
  * CNS1 status must be documented at time of screening by CSF assessment. Patients with prior CNS2 or CNS3 disease must be CNS1 at screening and have no residual CNS deficits or symptoms.
  * Patients will need to adhere to institutional contraception guidelines for a minimum of 1 year.

Exclusion Criteria:

* Concurrent active malignancy excluding non-melanoma skin cancer. Patients with a history of prior malignancy who have been treated with curative intent and have been in remission for at least 2 years are eligible.
* Burkitt's leukemia or lymphoma
* Patients with measurable extramedullary disease at screening are excluded. Patients with prior history of extramedullary disease are allowed after documentation of disease resolution by either PET/CT scan (or CT with contrast if PET cannot be performed).
* The following medications are excluded:

  * Steroids: Therapeutic doses of corticosteroids (greater than 10mg daily of prednisone or its equivalent) within 7 days of leukapheresis or 72 hours prior to CAR T cell infusion.
  * Systemic chemotherapy: Must be discontinued 7 days prior to leukapheresis or 7 days prior to starting lymphodepleting chemotherapy if used during bridging.
  * Tyrosine kinase inhibitors: Must be discontinued 48 hours prior to apheresis and 48 hours prior to starting lymphodepleting chemotherapy, if used during bridging.
  * Blinatumomab must be discontinued 5 days before apheresis
  * Inotuzumab must be discontinued 2 weeks before apheresis to allow T cell recovery
* Patients with uncontrolled systemic fungal, bacterial, viral or other infection at time of leukapheresis or at time of CAR T cell infusion
* Blinatumomab may not be used as bridging therapy following apheresis
* Positive test indicating the presence of active infection with the following pathogens: HIV, Hepatitis B (detectable Hep B DNA by PCR or Hep B surface antigen), Hepatitis C (detectable Hep C RNA by PCR), HTLV, Syphilis. The tests required will be agreed upon with the manufacturer to comply with manufacturer's regulatory and manufacturing requirements.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
relapse free survival (RFS) (Cohort A) | 1 year from infusion
  The time from CAR T infusion until non-response, relapse, or death of any cause, censored at last follow up. Non-response will be defined as the presence of > 5% abnormal lymphoblasts in the bone marrow, or the presence of unequivocal CNS or extramedullary disease after obe-cel infusion. Relapse will be defined as the emergence of > 5% abnormal lymphoblasts in the bone marrow, or the emergence of new unequivocal CNS or extramedullary disease after obe-cel infusion. Patients will be censored for relapse free survival if they undergo allogenic stem cell transplant or receive any other new treatment (except start or change of TKI maintenance) while in remission.

SECONDARY OUTCOMES:
Minimal residual disease (MRD)-negative Event Free Survival (EFS) (Cohort A & B) | 1 year from infusion
  The time from CAR T infusion until non-response (including MRD), relapse (including MRD), or death of any cause, censored at last follow up. MRD will be measured in the bone marrow as described above and considered positive if >10-^4.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack - Suffolk (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/